CLINICAL TRIAL: NCT01831570
Title: Prospective 6 Years Follow up of Patients With Hand Osteoarthritis
Brief Title: DIGItal Cohort Osteoarthritis Design
Acronym: DIGICOD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K110301
Record Dates: First submitted 2013-03-29; First posted 2013-04-15 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Arthrosis of Hand
Keywords: Hand osteoarthritis; predictive factors; erosive hand OA
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- symptomatic and radiographic hand osteoarthritis (Other): Patients above 35-years old with symptomatic and radiographic hand osteoarthritis
  Interventions: Other: GENETIC and radiographs

INTERVENTIONS:
Other: GENETIC and radiographs — GENETIC : Blood sample for genetic analysis will be performed at inclusion in order to built a DNA collection OTHER: Serum samples will be performed at inclusion M0, M36 and M72 for serum biomarkers assessment OTHER : These radiographs will be performed at M0, M36 and M72

SUMMARY:
Introduction Osteoarthritis is a chronic disease characterized by a progressive degradation of articular cartilage. Hand OA involves symptomatically more than 1 million of subjects in France (i.e., painful or with functional impairment). To date, the treatment of OA is only symptomatic and no drugs are able to stop the degradative process of cartilage.

50% of patients with hand OA exhibit a functional impairment responsible for a severe handicap, which is almost similar to rheumatoid arthritis. While the risk factors of hand OA are well identified (i.e., familial history, female sex, menopause, obesity), clinical outcome in large cohort is poorly known. In addition, the investigators miss predictive clinical, biological or imaging factors of severe clinical (i.e. pain, functional impairment or aesthetic damage) or structural evolution (i.e., aggravation of radiographic scores).

Primary objective To investigate in hand OA patients predictive clinical, biological, genetic and imaging factors of clinical aggravation after 6 years of follow-up.

Secondary objectives To investigate in hand OA patients predictive clinical, biological, genetic and imaging factors of clinical aggravation after 3 years of follow-up.

To investigate in hand OA patients predictive clinical, biological, genetic and imaging factors of clinical aggravation after 3 years of follow-up.

To investigate whether variations of clinical evaluation of hand hand OA and radiographic structural changes are associated or correlated between inclusion and 3 years of follow-up or between inclusion and 6 years follow-up To investigate whether clinical status and radiographic alterations are correlated at inclusion To determine whether hand OA is associated with OA at other sites or with other hand diseases (carpal tunnel syndrome, tendinitis) To evaluate frequency of erosive hand OA among the whole hand OA cohort at inclusion, at 3 and 6 years of follow-up To identify clinical, biological, genetic and imaging factors associated with erosive hand OA (versus non erosive hand OA) at inclusion or during the follow up (3 and 6 years) To investigate predictive clinical, biological, genetic and imaging factors of clinical or radiographic aggravation after 3 or 6 years of follow-up in the erosive hand OA subgroup

Methods :

the investigators plan to include 500 patients in the cohort (5/week) 7 visits (one per year) are planned: M0, M12, M24, M36, M48, M60 and M72. A clinical evaluation of hand OA will be performed at each visit. At visit M0, M36 and M72, hand radiographs and radiographs of other OA localisation (if symptomatic) will be performed.

A blood sample will be taken at inclusion for biomarker studies and genetic investigations.

A blood sample will be taken at M36 and M72 to build a prospective serum collection.

Duration of the study: 8.5 years with 2.5 years of inclusion period Duration of the study for one patient: 6 years Recruitment at the Rheumatology Department of Saint-Antoine Hospital with a multicentric international steering committee

Potential outcomes :

* Identification of clinical, radiological and biological tools useful to predict clinical and structural outcomes
* Description of the history course of hand OA and predictive factors of severe evolution (i.e. erosive form of hand OA) To integrate in daily practice, clinical and radiological tools allowing a standardized follow up of hand OA patients.

DETAILED DESCRIPTION:
Primary objective To investigate in hand OA patients predictive clinical, biological, genetic and imaging factors of clinical aggravation after 6 years of follow-up.

Secondary objectives To investigate in hand OA patients predictive clinical, biological, genetic and imaging factors of clinical aggravation after 3 years of follow-up.

To investigate in hand OA patients predictive clinical, biological, genetic and imaging factors of clinical aggravation between inclusion and 3 years of follow-up and between inclusion and the end of follow-up at 6 years.

To determine the clinical, biological and radiographic factors predictive of the radiographic progression of OA between inclusion and 3 years but also between inclusion and 6 years To investigate whether clinical changes and radiographic structural changes are associated or correlated between inclusion and 3 years of follow-up or between inclusion and 6 years of follow-up To investigate whether clinical status and radiographic alterations are correlated at inclusion To determine whether hand OA is associated with other OA at other sites or with other hand diseases (carpal tunnel syndrome, tendinitis) To evaluate frequency of erosive hand OA among the whole hand OA cohort at inclusion, at 3 and 6 years of follow-up To identify clinical, biological, genetic and imaging factors associated with erosive hand OA (versus non erosive hand OA) at inclusion or during the follow up (3 and 6 years) To investigate predictive clinical, biological, genetic and imaging factors of clinical or radiographic aggravation after 3 or 6 years of follow-up in the erosive hand OA subgroup To perform a cross-sectional analysis of the correlation between clinical tools and erosive radiographic involvement at inclusion (in the population with erosive hand OA at inclusion) ; To evaluate the frequency of fibromyalgia at 3 years of follow-up and at the end of the follow-up at 6 years ; To evaluate the frequency of neuropathic pain at 3 years of follow-up and at the end of the follow-up at 6 years ; To evaluate the pressure pain threshold at 3 years of follow-up and at the end of the follow-up at 6 years.

Methods : Prospective observational study The study will be proposed to all patients viewed at the out-patient clinic for hand OA which took place in Saint-Antoine Hospital in Rheumatology Department since 2004 (usually 12/week). The investigators plan to include 500 patients in the cohort (5/week).

7 visits (one per year) are planned: M0, M12, M24, M36, M48, M60 and M72. A clinical evaluation of hand OA will be performed at each visit. At visit M0, M36 and M72, hand radiographs and radiographs of other OA localisation (if symptomatic) will be performed.

A blood sample will be taken at inclusion for biomarker studies and genetic investigations.

A blood sample will be taken at M36 and M72 to build a prospective serum collection.

Duration of the study: 8.5 years with 2.5 years of inclusion period Duration of the study for one patient: 6 years Recruitment at the Rheumatology Department of Saint-Antoine Hospital with a multicentric international steering committee

ELIGIBILITY:
Inclusion Criteria:

* Patients above 35-years old, having hand OA according to one of the following definitions:
* symptomatic hand OA fulfilling ACR criteria on at least 2 joints among proximal interphalangeal, distal interphalangeal joints or 1st interphalangeal joint with Kellgren-Lawrence > 2
* symptomatic thumb base OA with Kellgren-Lawrence > 2

Exclusion Criteria:

* Inflammatory rheumatic destructive disorders (psoriatic arthritis, rheumatoid arthritis)
* Polyarthritis related to gout or chondrocalcinosis involving hand
* Secondary hand OA related to infection or traumatism
* Secondary OA related to genetic dysplasia
* Pregnancy and feeding

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Baseline clinical, biological, genetic and imaging factors of clinical aggravation after 3 years of follow-up(AUSCAN VA3.0) | 6 years
  Australian/Canadian Hand Osteoarthritis Index (AUSCAN VA3.0), Functional Index for Hand OA (FIHOA), modified short-form of Score for the Assessment and quantification of Chronic Rheumatic Affections of the Hands (M-Short Form-SACRAH), Arthritis Impact Measurement Scales (AIMS2), Health Questionnaire Assessment (HAQ), Hospital Anxiety and Depression Scale (HAD), Cochin index, Doyle index, synovial count, Heberden nodes count, Bouchard nodes count, grip strength, pinch strength, pain VAS, function VAS and aesthetic VAS at 6 years.

SECONDARY OUTCOMES:
Baseline clinical, biological, genetic and imaging factors of clinical aggravation after 3 years of follow-up(AUSCAN VA3.0) | 3 years
  association or correlation between clinical changes and radiographic structural changes between inclusion and 3 years of follow-up or between inclusion and 6 years of follow up
Kallman score, Verbruggen score, Kellgren-Lawrence grading and OARSI scoring (Altman score) | 3 and 6 years
patients above 35 years old with symptomatic and radiographic hand osteoarthritis | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis Berenbaum, PU PH, Principal Investigator — Assistance publique
Locations (1):
- Service de Rhumatologie - Hôpital Saint-Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cambon-Binder A, Jaisson S, Tuffet S, Courties A, Eymard F, Okwieka A, Gillery P, Miquel A, Rousseau A, Crema MD, Berenbaum F, Sellam J. Serum carboxymethyllysine concentration is associated with erosive hand osteoarthritis. Osteoarthritis Cartilage. 2023 Jul;31(7):976-984. doi: 10.1016/j.joca.2023.03.006. Epub 2023 Mar 15. PMID 36931384
- [Derived] Binvignat M, Pires G, Tchitchek N, Costantino F, Courties A, Klatzmann D, Butte AJ, Combe B, Dougados M, Richette P, Mariotti-Ferrandiz E, Berenbaum F, Sellam J. Identification of Symptom Phenotypes of Hand Osteoarthritis Using Hierarchical Clustering: Results From the DIGICOD Cohort. Arthritis Care Res (Hoboken). 2023 Jul;75(7):1494-1502. doi: 10.1002/acr.25047. Epub 2023 Jan 25. PMID 36263851